CLINICAL TRIAL: NCT03367897
Title: Bleeding Ulcer and Erosions Study "BLUE Study"
Acronym: BLUE
Status: Completed | Type: Observational
Sponsor: Ostfold Hospital Trust (Other)
Collaborators: University Hospital, Akershus (Other)
Responsible Party: Sponsor
Other Study IDs: 1319
Record Dates: First submitted 2016-10-10; First posted 2017-12-11 (Actual); Last update posted 2019-11-18 (Actual); Status verified 2019-11

CONDITIONS: Bacterial Infection Due to Helicobacter Pylori (H. Pylori); Peptic Ulcer; Bleeding Ulcer
Keywords: Helicobacter pylori; peptic ulcer; erosions; bleeding; Nsaids; Noac
MeSH Terms: conditions — Peptic Ulcer; Hemorrhage

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Bleeding ulcer/erosions: Patients with hematemesis and/or melena, anemia or positiv FOBT that during gastroscopy are diagnosed with ulcer and/or erosions of the ventricle and/or duodenum. Gastroscopy must be performed within 72 hours of the findings above.
- Peptic ulcer without bleeding: Control group for H. pylori will be patients with peptic ulcer without bleeding. These patients are systematically registered at SØ from August 2013 through the ongoing European registration study - HpEuReg study. SØ participate in this study, together with 9 other Norwegian hospitals, which is approved by REK.

SUMMARY:
A prospective study of bleeding peptic ulcers and/or erosions in the upper gastrointestinal tract - risk-medication, presence of Helicobacter pylori, treatment and outcome.

DETAILED DESCRIPTION:
Patients admitted to hospital due to hematemesis and/or melena with endoscopic finding of ulcer and/or erosion in the ventricle and/or duodenum are eligible for inclusion in the BLUE study after an informed consent has been obtained. The gastroscopy must be performed within 72 hours after admission. Epidemiological data, comorbidity and past clinical history are recorded in addition to the consumption of defined risk medication and proton-pump inhibitors (PPI) during the last 4 weeks.

The Forrest classification is used to describe an ulcer if present at endoscopy and endoscopic modalities for treatment are used according to established recommendations. Surgery or radiological intervention will be applied if needed.

An infection with H. Pylori is diagnosed by different methods including a rapid urease test, culture and serology. If one of these tests is positive, the patient will receive triple therapy. To secure successful eradication patients are tested with 13C UBT (breath test) or HP antigen stool test after 3 months and HP IgG serology after 6 months.

Registration of lowest haemoglobin (Hb) level during hospitalization and an algorithm to treatment with blood transfusion and/or high dose IV iron will be performed to evaluate alternative treatments to blood transfusions alone. Effect of treatment is evaluated at 8 weeks and 6 months. A follow-up gastroscopy and blood test is performed after 2-3 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years who consent to be enrolled in the study
* Patients with hematemesis and/or melena, anemia or positiv FOBT that during gastroscopy are diagnosed with ulcer and/or erosions of the ventricle and/or duodenum.
* Gastroscopy must be performed within 24 hours of the findings above.

Exclusion Criteria:

* Patients who do not wish to participate or are not competent to give consent.
* Patients that due to language problems or other reasons do not understand the content of the information about the study.
* Patients with erosions without hematemesis, in whom one diagnose possible bleeding source on colonoscopy.
* Patients with malignant ulcer, ulcer simplex or cameron lesions.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with hematemesis and/or melena, anemia or positiv FOBT that during gastroscopy are diagnosed with ulcer and/or erosions of the ventricle and/or duodenum. Gastroscopy must be performed within 24 hours of the findings above.
Sampling Method: Non-Probability Sample
Enrollment: 543 (Actual)
Dates: Start 2015-03 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2019-07 (Actual)

PRIMARY OUTCOMES:
Risk medication in peptic ulcer bleeding | 4 weeks
  Any use of NSAIDs (non-selective NSAIDs and / or COX-2 inhibitors), acetylsalicylic acid (ASA), other antiplatelet agents (non ASA antiplatelet agents), warfarin, DOAC, LMWH, H2 blockers and proton pump inhibitors during the last four weeks before the bleeding episode.

SECONDARY OUTCOMES:
PPI prophylaxis in in peptic ulcer bleeding | 4 weeks
  Any use of PPI inhibitors during the last four weeks before the bleeding episode.
H. pylori infection rate | 4 weeks
  Gastric biopsies: 2 from the antrum and 2 from the corpus for culture, 1 the antrum and 1 from the corpus for rapid urease test (BIOHIT).
  Blood test sampling for ELISA IgG anti-HP antibodies.
In vitro H. pylori resistance to antibiotics | 2 weeks
  In vitro metronidazole susceptibility testing
Eradication rate of H. pylori using OAM triple therapy | 6 months
  3 months: 13C UBT (breath test) or HP antigen stool test. 6 months: ELISA IgG anti-HP antibodies

OTHER OUTCOMES:
Long-term effect of blood transfusion versus treatment with high-dose intravenous iron. | 6 months
  Blood samples

CONTACTS AND LOCATIONS:
Overall Officials: Jørgen Jahnsen, prof MD PhD, Principal Investigator — Institute of Clinical Medicine, University of Oslo and Akershus University Hospital
Locations (2):
- Norway (2):
  - Akershus University Hospital, Oslo
  - Ostfold Hospital Trust, Sarpsborg, Østfold fylke

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Romstad KK, Thomas O, Soberg T, Detlie TE, Ricanek P, Jahnsen ME, Lerang F, Jahnsen J. High consumption of risk medication and underutilization of proton pump inhibitors among patients with upper gastrointestinal bleeding due to peptic ulcers and erosions (BLUE study). Scand J Gastroenterol. 2026 Jan;61(1):44-52. doi: 10.1080/00365521.2025.2594780. Epub 2025 Dec 16. PMID 41400236
- [Derived] Romstad KK, Detlie TE, Soberg T, Thomas O, Ricanek P, Jahnsen ME, Lerang F, Jahnsen J. Treatment and outcome of gastrointestinal bleeding due to peptic ulcers and erosions - (BLUE study). Scand J Gastroenterol. 2022 Jan;57(1):8-15. doi: 10.1080/00365521.2021.1988701. Epub 2021 Oct 18. PMID 34663154
- [Derived] Romstad KK, Detlie TE, Soberg T, Ricanek P, Jahnsen ME, Lerang F, Jahnsen J. Gastrointestinal bleeding due to peptic ulcers and erosions - a prospective observational study (BLUE study). Scand J Gastroenterol. 2020 Oct;55(10):1139-1145. doi: 10.1080/00365521.2020.1819405. Epub 2020 Sep 15. PMID 32931710